CLINICAL TRIAL: NCT00421265
Title: Prospective Cohort Study of Active Surveillance for Prostate Cancer With Indolent Linical Features
Brief Title: Active Surveillance for Prostate Cancer With Indolent Features
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 138/06
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; active surveillance; indolent features
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
In patients with prostate cancer with indolent features, disease progrssion may be very slow and in many cases will never become clinically evident during the patient's lifetime. Active surveillance is a continuous process of monitoring disease characteristcs aiming to avoid the morbidity of active therapy in patients with stabe indolent parameters, while offering early detection of disease activity in others who will need active therapy to control their disease. We hypothesize that active surveillance will permit the avoidance of therapy related morbidity in the majority of appropriate patients and will be associated with maintaining their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Men 65 years of age or older who were diagnosed with prostate cancer in the past 3 month prior to inclusion
2. Gleason's score of 6 or less.
3. Clinical T1C per digital rectal exam.
4. Pre biopsy PSA serum level of 6.0ng/ml or less.
5. The presence of cancer in a single biopsy core of at least 8 taken.
6. The presence of cancer in no more than 10% of the length of the core involved.
7. Patient's consent to engage in active surveillance after being informed of the benefits and potential risks of this approach as well as of alternative lines of therapy.
8. Israeli residence with the readiness to be available for the followup schedule.

Exclusion Criteria:

Patients who do not meet the above eligibility criteria

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150

CONTACTS AND LOCATIONS:
Overall Officials: Dan Leibovici, M.D., Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel